CLINICAL TRIAL: NCT06820840
Title: Comparative Clinical Performance of Hybrid Resin Composite vs. Hybrid Ceramic Onlays in the Restoration of Carious Molars: A Randomized Clinical Trial
Brief Title: Hybrid Resin Composite vs. Hybrid Ceramic Onlays for Restoring Carious Molars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peter Medhat Youssef Gerges (Other)
Responsible Party: Sponsor-Investigator, Peter Medhat Youssef Gerges, Assistant Lecturer - Conservative Dentistry Department - MIU, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PGCU-6-2-2025
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Carious Molars
Keywords: Onlay; Onlays; Hybrid resin composite; Hybrid ceramic; SHOFU; Ceramage; S-PRG; SPRG; Vital molars; Block HC Hard

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hybrid Ceramic Onlay (Active Comparator)
  Interventions: Other: SHOFU Block HC Hard
- Hybrid Resin Composite Onlay (Experimental)
  Interventions: Other: SHOFU Ceramage

INTERVENTIONS:
Other: SHOFU Block HC Hard — Cementation of hybrid ceramic onlay (SHOFU Block HC Hard) on carious molars.
  Arms: Hybrid Ceramic Onlay
Other: SHOFU Ceramage — Cementation of hybrid resin composite onlay (SHOFU Ceramage) on carious molars.
  Arms: Hybrid Resin Composite Onlay

SUMMARY:
The goal of this clinical trial is to compare the clinical performance of hybrid resin composite and hybrid ceramic onlays in restoring carious molars. It will also evaluate the wear resistance of both materials. The main questions it aims to answer are:

* Does the hybrid resin composite or hybrid ceramic onlay perform better in clinical settings over time?
* How much wear occurs in each type of onlay over 18 months?

Researchers will compare SHOFU Ceramage (hybrid resin composite) to SHOFU Block HC Hard(hybrid ceramic) to see which material performs better in restoring molars with extensive caries.

Participants will:

* Receive either a hybrid resin composite or hybrid ceramic onlay for their molar cavities.
* Visit the clinic for checkups at baseline, 6 months, 12 months, and 18 months.
* Undergo visual assessments of their restorations and quantitative wear analysis during follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Able to tolerate necessary restorative procedures
* Willing to sign the informed consent
* Accepts the follow-up period

Exclusion Criteria:

* ICDAS 4/5 cavities in first and second permanent molars
* Onlay cavities with at least one cusp coverage
* Patients with acceptable oral hygiene

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Clinical Performance | From baseline to 18 months
  Measured using modified USPHS criteria

SECONDARY OUTCOMES:
Quantitative Wear Analysis | From baseline to 18 months
  Measured in micrometers (μm) using a three-dimensional surface-based superimposition software

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (ICF) Clinical Study Report (CSR)
Supporting Information: Study Protocol, SAP, ICF, CSR